CLINICAL TRIAL: NCT00737516
Title: A Centralized Cord Blood Registry to Facilitate Allogeneic, Unrelated Donor Umbilical Cord Blood Transplantation
Brief Title: Centralized Cord Blood Registry to Facilitate Unrelated Cord Blood Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: T00004
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: Registry; Unrelated Umbilical Cord Blood donor; Hematopoietic Reconstitution; Center for Cord Blood; Bone Marrow Transplantation
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): HPC, Cord Blood
  Interventions: Biological: HPC, Cord Blood

INTERVENTIONS:
Biological: HPC, Cord Blood — Search for HLA compatible cord blood units using the NMDP registry

SUMMARY:
The National Marrow Donor Program (NMDP) has established a system for registering, matching, and tracking unrelated donor cord blood units (CBUs) and transplant outcomes. Study subjects are donors who enroll through collaborating cord blood banks. This study creates uniform collection, screening, testing and storage requirements for cord blood units. The purpose of standardization is to improve efficiency in the selection of cord blood units for transplantation.

DETAILED DESCRIPTION:
The NMDP Cord Blood registry is organized as a network of member cord blood banks and transplant centers whose interactions are managed by the NMDP's Center for Cord Blood. Banks agree to comply with uniform collection, screening, testing and storage requirements. Upon approval of membership, cord blood banks submit detailed information on each stored CBU for registration into a proprietary computer system. A transplant center, working on behalf of potential recipients, submits search requests to the NMDP and receives electronic reports detailing potentially suitable CBUs. From these reports, the transplant center selects a CBU(s) for further testing, which includes at a minimum confirmation of the CBUs Human Leukocyte Antigen (HLA) typing data. Upon final selection of the desired CBU for transplantation, arrangements are made for timely shipment of the unit to the transplant center. Following transplantation, recipient outcome data are submitted by the transplant center for addition to the study database.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3621 (Actual)
Dates: Start 2000-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Study safety and efficacy for treatment for malignant and non-malignant disorders | annually

SECONDARY OUTCOMES:
Study relationship between HLA disparity and survival | annually

CONTACTS AND LOCATIONS:
Overall Officials: John P Miller, M.D., Ph.D., Principal Investigator — National Marrow Donor Program
Locations (19):
- United States (19):
  - StemCyte International Cord Blood Center, Covina, California
  - Children's Hospital of Orange County Cord Blood Bank, Orange, California
  - Ashley Ross Cord Blood Program, San Diego, California
  - University of Colorado Cord Blood Bank, Aurora, Colorado
  - Bonfils Cord Blood Service, Denver, Colorado
  - Lifeforce Cryobanks, Altamonte Springs, Florida
  - Gift of Life Marrow Foundation, Boca Raton, Florida
  - LifeCord, Gainesville, Florida
  - ITxM Cord Blood Services, Glenview, Illinois
  - J.P. McMarthy Cord Stem Cell Bank, Detroit, Michigan
  - Michigan Community Blood Centers, Grand Rapids, Michigan
  - St. Louis Cord Blood Bank, St Louis, Missouri
  - CBS - New Jersey Cord Blood bank, Allendale, New Jersey
  - Coriell - New Jersey Cord Blood Bank, Camden, New Jersey
  - Carolinas Cord Blood Bank, Durham, North Carolina
  - Cleveland Cord Blood Center, Cleveland, Ohio
  - M.D. Anderson Cord Blood Bank, Houston, Texas
  - Texas Cord Blood Bank, San Antonio, Texas
  - Puget Sound Blood Center, Seattle, Washington